CLINICAL TRIAL: NCT03596918
Title: Longitudinal Quality of Life Study Among Participants With AIDS-Associated Kaposi Sarcoma at Bugando Medical Centre, in Mwanza, Tanzania
Brief Title: Evaluating Quality of Life in Patients With AIDS-Associated Kaposi Sarcoma Treated With Bleomycin and Vincristine
Status: Completed | Type: Observational
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry); University of Arkansas (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: AMC-S007; NCI-2017-01864 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AMC-S007 (Other: AIDS Malignancy Consortium); AMC-S007 (Other: CTEP); UM1CA121947 (NIH)
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Results first posted 2022-07-25 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: AIDS-Related Kaposi Sarcoma; Human Immunodeficiency Virus 1 Positive
MeSH Terms: conditions — AIDS-related Kaposi sarcoma | interventions — Bleomycin; Vincristine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Supportive care (vincristine sulfate, bleomycin sulfate): Patients receive vincristine sulfate IV over 1-2 minutes and bleomycin sulfate IV over 10 minutes on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bleomycin Sulfate; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Vincristine Sulfate

INTERVENTIONS:
Biological: Bleomycin Sulfate — Given IV
  Other Names: Blanoxan; BleMomycine; Blenoxane; Bleo-cell; Bleo-S; Bleocin; Bleolem; Bleomycin Sulfas; Bleomycin Sulphate; Blexane; Oil Bleo
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This pilot phase I trial studies how well treatment with vincristine and bleomycin affect quality of life in patients with acquired immunodeficiency syndrome (AIDS)-associated Kaposi sarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the longitudinal quality of life of participants with human immunodeficiency virus (HIV)-associated Kaposi sarcoma (KS) during treatment with bleomycin sulfate (bleomycin) and vincristine sulfate (vincristine) at a single institution in East Africa.

SECONDARY OBJECTIVES:

II. To explore baseline and time-dependent correlates of improvements in quality of life (QOL).

TERTIARY OBJECTIVES:

III. To assess quality control (completeness and accuracy) in data capture of adverse events, clinical benefit, and objective response for site evaluation and training purposes.

OUTLINE:

Patients receive vincristine intravenously (IV) over 1-2 minutes and bleomycin IV over 10 minutes on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 ribonucleic acid (RNA) viral load

  * NOTE: the term "licensed" refers to a United States (U.S.) FDA-approved kit or for sites located in countries other than the U.S., a kit that has been certified or licensed by an oversight body within that country and validated internally
  * World Health Organization (WHO) and Centers for Disease Control and Prevention (CDC) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment; a reactive initial rapid test should be confirmed by either another type of rapid assay or an E/CIA that is based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a Western blot or a plasma HIV-1 ribonucleic acid (RNA) viral load
* Participants must have pathologically confirmed Kaposi sarcoma
* Participants should not have had prior therapy for their Kaposi sarcoma
* All participants must be on stable antiretroviral therapy (ART) for a minimum of 12 weeks prior to study entry with an acceptable regimen that adheres to national guidelines for treatment of HIV infection
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky performance status >= 50%)
* Leukocytes: >= 3,000/mm^3, within 7 days of enrollment
* Absolute neutrophil count: >= 1,000/mm^3, within 7 days of enrollment
* Hemoglobin >= 8 g/dL, within 7 days of enrollment
* Platelets: >= 75,000/mm^3, within 7 days of enrollment
* Direct bilirubin: < 3 mg/dL, within 7 days of enrollment
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) / alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]): =< 2.5 x institutional upper limit of normal, within 7 days of enrollment
* Creatinine:

  * Creatinine levels within normal institutional limits, within 7 days of enrollment; or,
  * Creatinine clearance >= 60 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal, within 7 days of enrollment
* Participants with serious chronic, acute, or recurrent infections must have completed at least 14 days of therapy prior to study entry and be clinically stable
* If the participant is a female of childbearing potential (FCBP), defined as a sexually mature woman who: (1) has not undergone a hysterectomy or bilateral oophorectomy, or (2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months), the participant must have a negative urine or serum pregnancy test within 1 week prior to enrollment and agree to use an effective form of contraception (e.g., barrier contraception or hormonal contraception), during the 5 months of planned chemotherapy treatment and for 6 months after completing treatment
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who are receiving any other investigational agents
* Participants with known brain metastases
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to bleomycin or vincristine
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Participants who are breastfeeding a child; breastfeeding should be discontinued if the mother is treated with this chemotherapy
* Current or history of known pulmonary fibrosis, chronic obstructive pulmonary disease (COPD), emphysema, bronchiectasis, or diffuse or significant local radiographic interstitial infiltrates on chest x-ray (CXR) or computed axial tomography (CT) scan, that, in the opinion of the investigator, would exclude bleomycin use

  * NOTE: participants with an abnormal CXR or CT scan (which may indicate pulmonary KS) should undergo screening evaluations to rule out an infectious cause, per standard of care; if available, other diagnostic procedures such as bronchoscopy should be considered to confirm the presence or absence of pulmonary KS and/or an infectious agent; these procedures should be completed outside the study; these participants should be excluded if, in the opinion of the site investigator, use of bleomycin would be detrimental
* Oxygen saturation less than 90% and/or exercise desaturation greater than 4% within 14 days before study enrollment

  * NOTE: exercise is defined as any activity that will increase a participant?s resting heart rate by at least 20 beats/minute

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from the clinical care population presenting to Bugando Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-06-13 (Actual); Study Completion 2020-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Schroeder, Study Chair — AIDS Malignancy Consortium; Nestory Masalu, Study Chair — Bugando Medical Centre
Locations (1):
- Bugando Medical Centre, Mwanza, Tanzania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supportive Care (Vincristine Sulfate, Bleomycin Sulfate)
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Supportive Care (Vincristine Sulfate, Bleomycin Sulfate)
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (16.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Tanzania | 10

OUTCOME MEASURES:

1. Primary Outcome: Total Score on Quality of Life Assessed Using Functional Assessment of Cancer Therapy-General (FACT-G) Questionnaire
Description: The four domains of the FACT-G questionnaire will be determined for each questionnaire: physical well-being, social/family well-being, emotional well-being, and functional well-being. Each of these four domains is scored on a subset of 6-7 statements with a 0-4 scale. The domain is scored by summing up the responses to these statements. The ranges for the domains are as follows: physical well-being 0-28, social/family well-being 0-28, emotional well-being 0-24, and functional well-being 0-28. Using general estimating equations, changes in these domains with time will be explored. Logistic regression analyses will be used to correlate changes in quality of life domains with clinical response.
  The overall score is the sum of all the subscales and ranges from 0 to 108. Higher scores reflect better quality of life outcomes.
  The FACT-G Total Score at 3 months is reported here
Time Frame: Up to 3 months after treatment completion
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Supportive Care (Vincristine Sulfate, Bleomycin Sulfate)
Number analyzed (Participants) | 10
score on a scale | 56.9 (11.7)

2. Other Pre Specified Outcome: Clinical Data Collection Quality for Site Evaluation and Training Purposes
Description: Longitudinal Quality of Life Study Among Participants with AIDS-Associated Kaposi Sarcoma at Bugando Medical Centre, in Mwanza, Tanzania
Time Frame: Up to 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Supportive Care (Vincristine Sulfate, Bleomycin Sulfate)
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT03596918/Prot_SAP_000.pdf